CLINICAL TRIAL: NCT03047083
Title: Treatment Patterns and Key Healthcare Resource Use in Acute Myeloid Leukemia With and Without FLT3 Mutation
Brief Title: Treatment Patterns and Key Healthcare Resource Use in Acute Myeloid Leukemia (AML) With or Without FMS-like Tyrosine Kinase-3 (FLT3) Mutation Study Based on Retrospective Chart Review
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2215-MA-3074
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Retrospective; Non-interventional Study; FMS-like tyrosine kinase-3 (FLT3) mutations
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- IC eligible AML patients with FLT3 mutation: Newly diagnosed AML patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources
- IC ineligible patients with FLT3 mutation: Newly diagnosed AML patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources
- AML patients after R/R with FLT3 mutation: R/R are relapse/refractory patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources
- IC eligible patients without FLT3 mutation: Newly diagnosed AML patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources
- IC ineligible patients without FLT3 mutation: Newly diagnosed AML patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources
- AML patients after R/R without FLT3 mutation: R/R are relapse/refractory patients
  Interventions: Other: Treatment patterns among AML patients; Other: AML-related healthcare resources

INTERVENTIONS:
Other: Treatment patterns among AML patients — This is a retrospective cohort study of AML patients with or without FLT3 mutation who were exposed to treatments for AML per treating physician's decision between 1 January 2013 and 31 December 2015.
Other: AML-related healthcare resources — This is a retrospective cohort study of AML patients with or without FLT3 mutation who were exposed to treatments for AML per treating physician's decision between 1 January 2013 and 31 December 2015.

SUMMARY:
The purpose of this study is to retrospectively evaluate the treatment patterns and AML-related key healthcare resource use among AML patients, stratified by FLT3 mutation status, intensive chemotherapy (IC) eligibility, and relapsed or refractory (R/R) status.

DETAILED DESCRIPTION:
The current study is a retrospective non-interventional study using real-world data collected from existing medical records to evaluate descriptively the treatment patterns and key healthcare resource use among AML patients with or without FLT3 mutation. The current study relies on secondary use of existing data, and there is no intervention involved. Patients who received the first AML treatment after the initial diagnosis, or were classified as relapsed/refractory (R/R), between January 1, 2013 and December 31, 2015 will be randomly selected to be included in this study, and the data from their existing medical records will be extracted. Eligible patients will be grouped based on FLT3 mutation status, intensive chemotherapy (IC) eligibility, and R/R status.

For newly diagnosed patients, the index date will be defined as the initiation date of the first AML treatment following initial diagnosis. For the R/R patients, the index date will be defined as the date of the patient being classified as R/R. The study period will be the period from the index date to last follow-up date or death, whichever comes earlier. The endpoint measurements of this study are treatment patterns and key AML-related healthcare resources used during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML but NOT acute promyelocytic leukemia (APL)
* Known FLT3 mutation status
* Under the care of the participating physician during the past 3 years OR from the initial diagnosis of AML
* The medical records related to AML for the patient are available to the physician and can be abstracted for this study
* The medical records contains complete information on treatments and AML-related hospitalization, including admission date, length of stay, and reason of hospitalization
* Initiation date of first treatment after AML diagnosis OR date of being classified as relapsed from or being refractory to initial treatment (R/R) is between January 1, 2013 and December 31, 2015

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AML patients with or without FLT3 mutation under or previously under the care of participating physicians.
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

PRIMARY OUTCOMES:
Treatment patterns assessed by drugs initiated | Up to 3 years
Treatment patterns assessed by dosage | Up to 3 years
Treatment patterns assessed by duration of treatment | Up to 3 years
Treatment patterns assessed by whether remission was achieved. | Up to 3 years
Treatment patterns assessed by an event | Up to 3 years
  Reported death, failure of treatment or relapse of any type
AML-related healthcare resource use assessed by number of hospitalizations and lengths of ICU hospital stay | Up to 3 years
AML-related healthcare resource use assessed by number of emergency department (ED) visits | Up to 3 years
AML-related healthcare resource use assessed by number of outpatient visits | Up to 3 years
AML-related healthcare resource use assessed by number of blood transfusions | Up to 3 years
AML-related healthcare resource use assessed by number of infections and associated treatments | Up to 3 years
AML-related healthcare resource use assessed by number of lab tests | Up to 3 years
  Lab tests include bone marrow biopsy
AML-related healthcare resource use assessed by number of relevant concomitant medications | Up to 3 years
AML-related healthcare resource use assessed by number of diagnostic procedures | Up to 3 years
AML-related healthcare resource use assessed by use of mechanical ventilation | Up to 3 years
AML-related healthcare resource use assessed by use of parenteral feeding | Up to 3 years
AML-related healthcare resource use assessed by length of hospice care | Up to 3 years
AML-related healthcare resource use assessed by number of hospitalizations (ICU and non-ICU) | Up to 3 years
AML-related healthcare resource use assessed by lengths of hospital stay (ICU and non-ICU) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Medical Affairs, Global, Study Director — Astellas Medical Affairs, Global
Locations (1):
- Sermo, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.